CLINICAL TRIAL: NCT03394196
Title: Implementation and Evaluation of an HIV-2 Viral Load and ARV Resistance Informed Algorithm for 2nd-line ART in HIV-2 Infected Patients in the Initiative Sénégalaise d'Accès Aux Antirétroviraux (ISAARV) Program
Brief Title: RESIST-2: 2nd-line ART for HIV-2 Infection
Acronym: RESIST-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 and Funding
Sponsor: University of Washington (Other)
Collaborators: Clinique des Maladies Infectieuses, CHNU de Fann, Dakar, Senegal (Unknown); Centre de Sante de Ziguinchor, Casamance, Senegal (Unknown); Janssen Pharmaceutica (Industry); Merck Sharp & Dohme LLC (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Geoffrey S. Gottlieb, Professor, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000228; R01AI120765 (NIH)
Record Dates: First submitted 2017-12-14; First posted 2018-01-09 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: HIV-2 Infection
MeSH Terms: interventions — Zidovudine; BID protein, human; Lamivudine; Tenofovir; Emtricitabine; Lopinavir; Ritonavir; Raltegravir Potassium; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No HIV-2 resistance (Experimental)
  Interventions: Diagnostic Test: HIV-2 Genotypic Drug Resistance Testing using DBS; Drug: 2nd line ART ( Zidovudine 300mg BID + Lamivudine 150mg BID or Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID)
- HIV-2 NRTI resistance only (Experimental)
  Interventions: Diagnostic Test: HIV-2 Genotypic Drug Resistance Testing using DBS; Drug: 2nd line ART (Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID + Raltegravir 400mg BID )
- HIV-2 NRTI and PI resistance (Experimental)
  Interventions: Diagnostic Test: HIV-2 Genotypic Drug Resistance Testing using DBS; Drug: 2nd line ART (Tenofovir DF 300mg QD + Lamividine 300mg QD or Tenofovir DF 300mg QD + Emtricitabine 200mg QD + Darunavir 600mg BID-Ritonavir 100mg BID +Raltegravir 400mg BID)

INTERVENTIONS:
Diagnostic Test: HIV-2 Genotypic Drug Resistance Testing using DBS — Real time HIV-2 genotypic drug resistance testing using dried blood spots and consensus sequencing.
Drug: 2nd line ART ( Zidovudine 300mg BID + Lamivudine 150mg BID or Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID) — 1. No resistance: Continue Current ART: Zidovudine 300mg BID + Lamivudine 150mg BID or Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID (AZT/3TC or TDF/3TC or TDF/FTC + LPV/r) + Enhanced Adherence Counseling
  Arms: No HIV-2 resistance
Drug: 2nd line ART (Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID + Raltegravir 400mg BID ) — 2. NRTI resistance only: Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID + Raltegravir 400mg BID (TDF/FTC or TDF/3TC + LPV/r + RAL) + Enhanced Adherence Counseling
  Arms: HIV-2 NRTI resistance only
Drug: 2nd line ART (Tenofovir DF 300mg QD + Lamividine 300mg QD or Tenofovir DF 300mg QD + Emtricitabine 200mg QD + Darunavir 600mg BID-Ritonavir 100mg BID +Raltegravir 400mg BID) — 3. NRTI-PI resistance: Tenofovir DF 300mg QD + Lamividine 300mg QD or Tenofovir DF 300mg QD + Emtricitabine 200mg QD + Darunavir 600mg BID-Ritonavir 100mg BID +Raltegravir 400mg BID (TDF/FTC or TDF/3TC +DRV/r2 + RAL) + Enhanced Adherence Counseling
  Arms: HIV-2 NRTI and PI resistance

SUMMARY:
Prospective, longitudinal, open label, HIV-2 viral load and antiretroviral resistance informed 2nd-line ARV implementation study.

DETAILED DESCRIPTION:
Prospective, longitudinal, open label, HIV-2 viral load and antiretroviral resistance informed 2nd-line ARV implementation study.

DURATION

Up to 3 years

SAMPLE SIZE

150

POPULATION

HIV-2-infected adults (≥18 years old); ARV-experienced, with virologic failure on 1st-line 2NRTI+LPV/r in the ISAARV program.

STRATIFICATION

By ARV resistance

REGIMEN OR INTERVENTION

Intervention: Implement real time ARV resistance testing using rapid DBS/CS ARV Regimens: Based on ARV resistance testing

1. No resistance: Current ART: Zidovudine 300mg BID + Lamivudine 150mg BID or Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID (AZT/3TC or TDF/3TC or TDF/FTC + LPV/r) +Enhanced Adherence Counseling
2. NRTI resistance only: Tenofovir DF 300mg QD + Lamividine 300mg QD or Emtricitabine 200mg QD + Lopinavir/Ritonavir 400/100mg BID + Raltegravir 400mg BID (TDF/FTC or TDF/3TC + LPV/r + RAL) + Enhanced Adherence Counseling
3. NRTI-PI resistance: Tenofovir DF 300mg QD + Lamividine 300mg QD or Tenofovir DF 300mg QD + Emtricitabine 200mg QD + Darunavir 600mg BID-Ritonavir 100mg BID + Raltegravir 400mg BID (TDF/FTC or TDF/3TC +DRV/r2 + RAL) + Enhanced Adherence Counseling

ELIGIBILITY:
Inclusion Criteria:

1. HIV-2 infection: confirmed by Determine (Alere, Inc.) & Immunocomb II (Alere, Inc.) or equivalent
2. Failing 1st line antiretroviral therapy (e.g. AZT/3TC or TDF/XTC + LPV/r; previous 3 NRTI or 2 NRTI regimens; previous Indinavir (IDV) use, current or previous Atazanavir (ATV) use; previous NNRTI use)
3. For females of reproductive potential: negative serum or urine pregnancy test
4. Men and women age >/=18 years
5. Ability and willingness of subject to provide informed consent

Exclusion Criteria:

1. HIV-1 or HIV-1/HIV-2 dual infection
2. Pregnancy or Breast-feeding
3. Lab Abnormalities

   * AST/ALT >2.5 X ULN
   * CrCl <30
4. Current or previous use of Integrase Inhibitors or Darunavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Death | up to 3 years
  all cause mortality
Loss to follow up | 1 year
  no contact with study for 1 year
Virologic Failure on 2nd line ART | up to 3 years
  VL >250 copies/ml
HIV-2 ARV resistance on 2nd line ART | up to 3 years
  by DBS genotyping

SECONDARY OUTCOMES:
New WHO stage 3 or 4 event > 6 months after starting ART | up to 3 years
  BY WHO criteria
Grade 3 or 4 adverse events | up to 3 years
  DAIDS definitions
CD4 T-cell count trajectory | up to 3 year after starting 2nd-line ART
  delta CD4 count per year

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey S Gottlieb, MD PhD, Principal Investigator — University of Washington
Locations (2):
- Senegal (2):
  - Centre de Sante de Ziguinchor, Ziguinchor, Casamance
  - Clinique des Maladies Infectieuses Ibrahima DIOP Mar/CRCF, Centre Hospitalier Universitaire de Fann, Dakar

IPD SHARING:
Plan to Share IPD: Yes
IPD shared on request with ORB approval on final cleaned dataset
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at end of study
Access Criteria: IRB approval

REFERENCES:
- [Derived] Raugi DN, Diallo K, Diallo MB, Faye D, Cisse O, Smith RA, Sall F, Sall EHI, Faye K, Diatta JP, Diaw B, Sambou J, Malomar JJ, Hawes SE, Seydi M, Gottlieb GS; University of Washington-Senegal HIV-2 Study Group. Resource and infrastructure challenges on the RESIST-2 Trial: an implementation study of drug resistance genotype-based algorithmic ART switches in HIV-2-infected adults in Senegal. Trials. 2021 Dec 18;22(1):931. doi: 10.1186/s13063-021-05902-5. PMID 34922614